CLINICAL TRIAL: NCT05480072
Title: Investigating the Effects of Palmitoylethanolamide (PEA) on Stress, Craving and Pain in Opioid Use Disorder
Brief Title: Endocannabinoids, Stress, Craving And Pain Effects Study
Acronym: ESCAPE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Primavera A. Spagnolo, MD, PhD, Assistant Professor/Research Scientist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P001440
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
Keywords: palmitoylethanolamide; stress; craving; pain
MeSH Terms: conditions — Opioid-Related Disorders; Pain | interventions — palmidrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEA 600 mg (Active Comparator): PEA capsules (600 mg twice a day) will be administered for 21 days
  Interventions: Drug: Palmitoylethanolamide
- Placebo (Placebo Comparator): Placebo capsules (600 mg twice a day) will be administered for 21 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Palmitoylethanolamide — Palmitoyethanolamide (PEA) s a dietary supplement with anti-inflammatory and analgesic properties. Subjects will receive PEA (Levagen+) 600 capsules mg twice daily (BID) orally from Day 1 to Day 21
  Other Names: Levagen+
  Arms: PEA 600 mg
Other: Placebo — Participants will receive placebo matched to 600 mg PEA (Levagen+) capsules BID orally from Day 1 to Day 21
  Arms: Placebo

SUMMARY:
Opioid use disorder (OUD) represents one of the most severe public health crises, with more than 2 million individuals affected in the United States. Existing treatments do not target and restore several key alterations triggering opioid craving and relapse, including increased response to stress, mood disturbances and greater sensitivity to pain, which are caused by prolonged exposure to opioids. This double-blind, randomized, placebo-controlled study will investigate the effects that palmitoylethanolamide (PEA), an endogenous molecule part of the endocannabinoid system available as a dietary supplement, exerts on these alterations and their underlying mechanisms, with the goal of identifying a novel therapeutic approach to reduce craving and prevent relapse in patients with OUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* DSM-5 diagnosis of OUD
* English speaking
* Receiving either buprenorphine or methadone for treatment of opioid use disorder for at least 3 consecutive months prior to enrollment
* Receiving a stable dose of buprenorphine or methadone for the duration of the study
* Agreeable to abstaining from using any cannabis or CBD products two weeks prior to enrollment in the study, and for the duration of the trial
* For women of childbearing potential: agreeable to use one of the following:

  * hormonal methods, such as birth control pills, patches, injections, vaginal rings, or implants
  * barrier methods (such as a condom or diaphragm) used with a spermicide (a foam, cream, or gel that kills sperm)
  * intrauterine device (IUD)
  * abstinence (no sex)

Exclusion Criteria:

* DSM-5 diagnosis of moderate-to-severe cannabis use disorder, alcohol use disorder, and/or psychostimulant use disorder [medical record review and health history form]
* Active, recurrent substance use within the last 3 months that will interfere with study participation and completion of study procedures [medical record review and health history form]
* History of psychotic, bipolar and schizoaffective disorders [medical record review and health history form]
* Lifetime psychiatric hospitalization or suicide attempt, as assessed by the health history form
* Recent history (within 2 years) of major depressive disorder [health history form and clinical interview]
* Currently pregnant or breastfeeding (female only) [pregnancy test/ self-reported]
* History of autoimmune or chronic inflammatory diseases [health history form] Current use of medications known to alter inflammatory and immune response [health history form] Raynaud's disease [health history form]
* BMI >45
* Hepatic liver enzymes greater than 3x upper normal limit
* Vital signs: HR ≤60 or ≥100, SBP ≤90 or ≥160, DBP ≤50 or ≥100, RR < 12 or > 20
* Recent history of clinically significant medical conditions including, but not limited to, malignancy (and treatment for malignancy), HIV, immunological, endocrine (including uncontrolled diabetes or thyroid disease), renal, GI, or hematological abnormalities that are uncontrolled* [health history form and medical record review]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
stress-induced opioid craving visual analog scale (VAS) | day 21
  decrease from baseline in experimentally-provoked stress-induced craving ratings as measured via the visual analog scale (0= no craving to 100= extremely strong craving). Lower scores indicate reduced craving

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided